CLINICAL TRIAL: NCT00143052
Title: Body Composition, Insulin Concentration, Androgens and Bone Status in Women Referred With Hirsutism
Brief Title: Bone Status and Insulin Resistance in Hirsutism
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Odense University Hospital
Other Study IDs: 003
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2008-06-24 (Estimated); Status verified 2008-06

CONDITIONS: Hirsutism
Keywords: Hirsutism; Bone status; Androgens; insulin
MeSH Terms: conditions — Hirsutism; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to investigate how the bones of hirsute women are different from bones of healthy women. The change in hormone content in the blood will also be investigated. The study can be used to evaluate whether it will be relevant to bone scan all newly referred hirsute women.

Hirsute women are often over-weight and often have an increased amount of the male sex hormone in their blood. Their blood tests often show changes reminding of the ones seen in diabetic patients.

All hirsute women referred to the department will undergo an investigation revealing the reason for the increased hair growth. The investigation includes clinical investigation (height, weight and degree of hair growth), blood tests (for hormone status and bone status analysis) and bone scanning of the abdomen (body composition).

The trial includes a group of 50 strongly hairy women and a control group of 50 healthy women with normal hair growth. They are matched by body weight, since weight has great importance for the bone mineral content and thereby for osteoporosis in the long run.

ELIGIBILITY:
Inclusion Criteria:

Hirsute subjects:

* Belonging to group 1 or 2.
* Age: 20-46
* Hirsute score: >7
* Written informed consent

Control group:

* Age: 20-46
* Hirsute score: 0 (without razing)
* Regular menses
* Written informed consent

Exclusion Criteria:

* Previous cosmetic treatment for hirsutism.
* Use of contraceptive pill (within the past 6 months)
* Systemic steroid treatment > 6 weeks (ever)
* Age above 46 years/post menopause (increased FSH)
* Recognized diabetes mellitus or other endocrine disease
* Eating disorder
* Serious, treatment demanding disease

Ages: 20 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: hirsute patients vs. controls
Enrollment: 50 (Actual)
Dates: Start 2002-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Glintborg, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Diabetes Research Center, Odense, Funen, Denmark